CLINICAL TRIAL: NCT05250232
Title: One Year Clinical Evaluation of Conservative Versus Conventional Ceramic Onlays
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, howaida ahmed el-hagrasy, assistant lereture must university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: resala
Record Dates: First submitted 2022-01-09; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- onlays conservative (Experimental): conservative onlays preparation with partial cusp coverage only defective cusps
  Interventions: Other: onlays conservative
- onlays conventional (Active Comparator): onlays preparation design conventional as all cusps covered with shoulder finish line preparation
  Interventions: Other: onlays conventional

INTERVENTIONS:
Other: onlays conservative — Partial coverage of cusps with shoulder finish line
  Arms: onlays conservative
Other: onlays conventional — all coverage of cusps as overlay with shoulder finish line
  Arms: onlays conventional

SUMMARY:
the aim of present study is to evaluate clinically the fracture liability , marginal adaptation , and patient satisfaction of conservative versus conventional ceramic Onlays use e-max press to restore defective restored molar with old restoration or caries. with one or more cusp defect

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria:

All subjects are required to be:

1-From 18-50 years old, be able to read and sign the informed consent document. 2- Have no active periodontal or pulpal diseases, have teeth with good restorations 3- Psychologically and physically able to withstand conventional dental procedures 4- Patients with teeth problems indicated for onlay restoration:

1. Decayed teeth
2. Teeth restored with defected filling restorations
3. Teeth with occlusal defect 5- Able to return for follow-up examinations and evaluation Exclusion criteria

   1. Patient less than 18 or more than 50 years
   2. Patient with active resistant periodontal diseases
   3. Patients with poor oral hygiene and uncooperative patients
   4. Pregnant women
   5. Patients in the growth stage with partially erupted teeth
   6. Psychiatric problems or unrealistic expectations
   7. Lack of opposing dentition in the area of interest

      -

      -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-02-27 (Estimated); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
evaluation of fracture resistance | one year
  fracture resistance of restorations postoperatively: assessment of the restoration for fracture resistance , by using Measuring device Modified United States Public Health Service (MUSPHS) parameters were used to compare the restorations at baseline and final examination use explorer Measuring unit .Discrete(scores)
  1. alpha no evidence of fracture
  2. bravo evidence of fracture

SECONDARY OUTCOMES:
evaluation of marginal adaptation | 1 year
  marginal adaptation of restorations postoperatively assessment by Measuring device Modified USPHS Criteria Measuring unit .Discrete(scores) use explorer
  1. alpha no visible evidence of ditching along the margin
  2. bravo visible evidence of ditching along the margin not extending to the DE junction
  3. charlie mismatch between restoration and tooth structure within the normal range of color, shade ,translucency
evaluation of patient satisfaction to the onlay restoration through questioning the patient about pain during eating , acceptability ,sensitivity | 1 year
  patient satisfaction of restoration use Questionnaire VAS* Measuring device Measuring unit Numerical(discrete) ('0' unsatisfied-'10' satisfied)

IPD SHARING:
Plan to Share IPD: Undecided